CLINICAL TRIAL: NCT06719804
Title: The Safety and Efficacy Evaluation of Propranolol as an Adjunctive Treatment for Focal Refractory Epilepsy: A Pilot Study
Brief Title: Propranolol Adjuvant Treatment of Focal Refractory Epilepsy (PATFRE)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-260-002
Record Dates: First submitted 2024-12-01; First posted 2024-12-06 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Epilepsy, Drug Resistant
Keywords: Propranolol; Focal Refractory Epilepsy; CAMP-PKA-MEK/ERK pathway; non-selective beta-adrenergic antagonists
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label single arm, drug propanolol (Experimental): All subjects will receive the experimental drug
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Oral administration is given solely for the epilepsy seizure event. Dosage: 20mg per dose; The patient's blood pressure and heart rate are monitored after the seizure; if the SBP is above 90 mmHg and the heart rate is above 60 beats per minute, then patients are instructed to take propranolol within 1 hour of a seizure . If the seizure frequency is excessively high, the interval between doses should be no less than 6 hours and the medication should not be administered more than 3 times a day.

SUMMARY:
The aim of this study is to evaluate the clinical efficacy of propranolol as an adjunctive treatment for refractory epilepsy. The significance of this research lies in exploring whether propranolol, as an inhibitor of the CAMP-PKA-MEK/ERK pathway, can provide anticonvulsant effects for a wider range of refractory epilepsy patients. The study holds the potential to offer a novel adjunctive anticonvulsant treatment strategy targeting the CAMP-PKA-MEK/ERK pathway, specifically administered for seizure events, and applicable to various forms of refractory epilepsy.

DETAILED DESCRIPTION:
Propranolol is a non-selective β-adrenergic receptor antagonist that blocks β1 and β2 adrenergic receptors, antagonizing sympathetic nervous stimulation and catecholamine effects. It is widely used in the treatment of various cardiovascular diseases. Additionally, propranolol can intervene in the reconsolidation process of pathological memories and is used to treat neuropsychiatric disorders such as post-traumatic stress disorder (PTSD) and drug addiction. Professor Huang Zhuo's team, using a conditioned epilepsy memory mouse model, administered propranolol during the "epilepsy memory" reconsolidation window (within 5 minutes) to inhibit the ERK pathway, significantly reducing subsequent seizure episodes induced by sensory stimuli. However, intervention outside the reconsolidation window (9 hours later) had no significant effect. This study, however, only verified the alleviating effect of propranolol treatment on subsequent seizures in an animal model, and its clinical efficacy in controlling epilepsy still needs further validation.

Based on the "epilepsy memory" mechanism, propranolol combined with memory recall reconsolidation paradigms is expected to become an effective adjunctive treatment for refractory epilepsy. Evaluating its efficacy and safety not only helps determine its therapeutic value in epilepsy treatment but also provides important guidance for clinical practice, playing a crucial role in the translation from basic research to clinical application.

Current small-sample animal studies have confirmed that administering propranolol within the "epilepsy memory" reconsolidation window can reduce the frequency of seizures and shorten the duration of seizures in epileptic mice. However, there is no large-scale clinical study validating the impact of propranolol on clinical seizures in patients. This study is a prospective, single-arm open-label trial aimed at preliminarily exploring the efficacy and safety of propranolol in the treatment of refractory epilepsy. The primary outcome measures are the proportion of patients with a ≥50% reduction in the frequency of refractory epilepsy seizures and a ≥50% reduction in epileptiform discharges on vEEG monitoring compared to baseline. Secondary outcomes include the severity of seizures (measured by the Liverpool Epilepsy Severity Scale) and the patient's quality of life (measured by the QOLIE-31-P scale). Adverse events during propranolol treatment will also be recorded, providing an objective assessment of the side effects and complications of propranolol in the treatment of epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age.
* Meet the 2017 International League Against Epilepsy (ILAE) diagnostic criteria for for focal seizures or focal seizures progressing to bilateral tonic-clonic seizures.
* Diagnosed with refractory epilepsy, having used at least two AEDs without effectiveness for 2 years. No drug interaction between current AEDs and propranolol, and a stable dose for at least 12 weeks prior to enrollment.
* Seizure duration ≥1 minute, with accompanying sensory impairment.
* At least 6 focal seizures within the 12 weeks preceding enrollment.
* EEG or MRI/CT results within the past 2 years, confirming the diagnosis of focal epilepsy.
* The use of vagus nerve stimulation (VNS) and deep brain stimulation (DBS) is permitted, need to implant at least 5 months and stable for at least 12 weeks before enrollment.The parameters should keep unchanged until the end of the study.
* Informed consent signed.

Exclusion Criteria:

* Diagnosed with generalized or hereditary epilepsy with ion channel gene mutations
* Psychogenic non-epileptic seizures within 12 months;
* Treatable causes of epilepsy (such as metabolic disorders, toxicity, infections, space-occupying lesions, or identified genetic abnormalities)
* Patients with only non-motor focal seizures, as classified by the 2017 ILAE.
* Seizure clusters within the 12 months.
* Tonic-clonic status epilepticus within12 months.
* Free of major medical illnesses including:
* Cardiac diseases (history of cardiac valve disease, coronary artery disease, congestive heart failure, A-V block, peripheral vascular disease, any cardiac arrhythmia/bradycardia)
* Histories of asthma, bronchospastic disease, or obstructive pulmonary disease
* Severe allergic reactions to medications which are included in the beta blocker family
* Currently treated with a beta adrenergic receptor antagonist or Previously used within 12 months
* Uncontrolled Diabetes (HbA1c of ≤ 8 if previously tested)
* Uncontrolled hypotension
* Immunodeficiency disorders, liver or kidney diseases, acute infections, or advanced-stage tumors.
* Participants with a history of medical conditions or surgeries that, in the investigator's judgment, could affect the absorption, distribution, or metabolism of the study drug (e.g., active peptic ulcers, ulcerative colitis, Crohn's disease, or bowel obstruction) or those with difficulty swallowing.
* Participants with any medical condition, mental health status, cognitive impairment, or intellectual disability that the investigator believes could increase the risk to the participant or interfere with their ability to participate in the clinical trial.
* Participants meeting any of the following laboratory criteria: alanine aminotransferase (ALT) >2× upper limit of normal (ULN), aspartate aminotransferase (AST) >2× ULN, alkaline phosphatase (ALP) >2× ULN, platelet count <80×10^9/L, neutrophil count <1.8×10^9/L, or creatinine clearance (CLcr) <30 mL/min (calculated by the Cockcroft-Gault formula).
* In the period of pregnancy, childbirth, lactation.
* Alcohol abuse or drug misuse within 2 years prior to medication.
* Participation in another clinical study within 3 months;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-05 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Seizure Frequency Per 28 Days | assessed per 28 days during the treatment.
  Percent change in 28-day frequency of seizures during the 40 week treatment and follow-up period relative to baseline
Seizure Responder Rate | short-term treatment period (ending at 3 months); long-term follow-up period (ending at 12 months).
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.

SECONDARY OUTCOMES:
Seizure Severity | Baseline observation period; short-term treatment period (ending at 3 months); long-term follow-up period (ending at 12 months).
  The percent change from baseline in seizure severity evaluated by Liverpool seizure severity scale (LSSS) .
Life quality evaluation | Baseline observation period; short-term treatment period (ending at 3 months); long-term follow-up period (ending at 12 months).
  Percentage change from baseline in Quality of Life in Epilepsy-31 inventory (QOLIE-31) score.
Adverse Events | through study completion, 12 months.
  Rate of adverse events which were judged to be study-related throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing; Zhuo Huang, PhD, Principal Investigator — Peking University School of Pharmaceutical Sciences

IPD SHARING:
Plan to Share IPD: No